CLINICAL TRIAL: NCT07191210
Title: A Co-Produced Comprehensive Transition Programme Designed Using Experience-Based Co-Design to Support First-Line Nurse Managers
Brief Title: Co-Designed Comprehensive Transition Programme for First-Line Nurse Managers
Acronym: CTP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Idoia Pardavila, PhD, Faculty of Nursing, University of Navarra, University of Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UNAV-CTP-2024; Chair of María Egea (Other Grant/Funding Number: University of Navarra)
Record Dates: First submitted 2025-09-09; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Transition to First-Line Nurse Manager Role
Keywords: Nursing leadership; First-line nurse managers; Nurse manager education; Mentorship; Leadership training; Co-Production

STUDY DESIGN:
Intervention Model Description: All participants will receive the Comprehensive Transition Programme (CTP), a multicomponent intervention including training sessions, mentorship, online learning, and reflective practice. No control or comparison group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Transition Programme (CTP) (Experimental): Participants will receive the Comprehensive Transition Programme (CTP), a multicomponent intervention including face-to-face training modules, online learning, mentorship, and reflective practice over a 3-month period.
  Interventions: Behavioral: Comprehensive Transition Programme (CTP)

INTERVENTIONS:
Behavioral: Comprehensive Transition Programme (CTP) — A co-designed, multicomponent educational programme delivered over three months to support nurses transitioning into first-line management roles. The programme integrates classroom training modules, online learning, mentorship by senior nurse managers, and structured reflective practice.

SUMMARY:
This study will pilot a Comprehensive Transition Programme (CTP) to support nurses who move into first-line nurse manager (FLNM) roles at Clínica Universidad de Navarra. The transition to frontline management can be challenging and is linked to uncertainty, workload stress, and role ambiguity. The CTP was co-designed with clinical nurses, FLNMs, nursing directors and chief nursing officers using experience-based co-design methods so that its content fits the organisation's practice model and priorities.

The programme combines classroom training, online learning, mentorship, and structured reflective practice. Participants complete brief assessments before and after the programme. The primary focus is to see whether leadership practices improve; we will also examine feasibility and acceptability to inform future refinement.

This pilot uses a simple pre-post design with data collected at baseline and immediately after the programme. Findings will be used to optimise the CTP and to guide broader implementation in the health system.

(Eligibility, outcomes, dates and intervention components are detailed in their specific sections of this record.)

DETAILED DESCRIPTION:
Rationale and aim. The move from bedside nursing to first-line nurse management is a critical career transition that requires new leadership, managerial and relational capabilities. In response, a multicomponent Comprehensive Transition Programme (CTP) was co-designed with stakeholders across organisational levels using experience-based co-design. The aim of this pilot is to generate preliminary evidence on usefulness and feasibility and to explore changes in leadership practices among novice FLNMs.

Design overview. Single-group, pre-post mixed-methods pilot conducted at a tertiary university hospital. Data are collected at two timepoints: baseline (prior to programme start) and immediately post-intervention. The primary outcome is change in leadership practices; additional indicators include acceptability, fidelity and qualitative insights from reflective narratives.

(Primary/secondary outcome measures, time frames and sample size appear in the Outcomes and Enrollment fields.)

Participants. Eligible participants are nurses on the institutional pathway to frontline management, including (a) clinical nurses with responsibility roles not yet formally appointed as supervisors; (b) FLNMs with <5 years' experience at the institution; and (c) FLNMs with prior experience elsewhere recently appointed at the institution. Participation is voluntary with written informed consent.

(Full inclusion/exclusion criteria are provided in the Eligibility section.)

Intervention (overview). The CTP is delivered over approximately three months and integrates:

Structured training on leadership and team management, care quality and improvement, communication, quality standards, and human resources/finance;

Mentorship by experienced nurse managers;

Online learning to reinforce key skills;

Reflective practice through guided narrative work and peer discussion. Delivery follows a common syllabus and mentoring framework to support consistency across participants.

(Specific components and any materials/providers are listed under Arms/Interventions.)

Implementation and fidelity. Standardised session objectives, shared teaching materials, common mentoring guidelines, and written instructions for reflective activities are used to promote consistency. Attendance and completion of activities are monitored as feasibility/fidelity indicators.

Data collection and analysis. Quantitative data are analysed descriptively and for pre-post change in leadership practices. Qualitative reflective narratives are appraised with a structured rubric and thematically analysed to capture perceived learning, role adjustment and relational practice. Integration of quantitative and qualitative strands supports interpretation of preliminary efficacy and feasibility.

(Instruments and time frames are specified in Outcome Measures.)

Ethics and data protection. The study has prior approval from the institutional Research Ethics Committee. All participants provide informed consent. Procedures follow applicable regulations for confidentiality and data protection.

Expected contribution. Results will inform refinements to content, sequencing and delivery of the CTP and support planning for a larger-scale evaluation and potential scale-up across services.

ELIGIBILITY:
Inclusion Criteria:

* Clinical nurses with responsibility roles at Clínica Universidad de Navarra (CUN) but not yet formally appointed as supervisors.
* First-Line Nurse Managers (FLNMs) with less than five years of managerial experience in the CUN.
* FLNMs with more than five years of managerial experience acquired mainly in other institutions but recently appointed as first-line managers at the CUN.
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Nurses with more than five years of continuous experience as FLNMs at the CUN.
* Nurses in middle or executive management roles (e.g., area directors, chief nursing officers).
* Clinical nurses without any responsibility or leadership role.
* Inability or unwillingness to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-03 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Change in leadership practices (Leadership Practices Inventory, LPI) | Up to 12 months (Baseline, 3 months, 6 months, 12 months)
  Leadership behaviours will be assessed using the Leadership Practices Inventory (LPI), a validated 30-item questionnaire covering five domains: Model the Way, Inspire a Shared Vision, Challenge the Process, Enable Others to Act, and Encourage the Heart. Scores range from 10 to 100 per domain, with higher scores indicating more frequent leadership behaviours. Mean change between baseline and post-intervention will be analysed.

SECONDARY OUTCOMES:
Quality of reflective narratives | Up to 12 months (Baseline, 3 months, 6 months, 12 months)
  Reflective narratives written by participants will be assessed using an evaluation tool adapted from the Nursing Professional Practice Model (NPPM-CUN). The tool evaluates three core managerial competencies-respect, intentional presence, and knowing the team-together with reflective capacity. Each item is rated on a 4-point scale (1 = not demonstrated, 4 = fully demonstrated). Mean scores and changes between baseline and post-intervention will be analysed, complemented with thematic analysis of narrative content.